CLINICAL TRIAL: NCT00580788
Title: Determining the Maximal Safe Dose of a Continuous Infusion of Parathyroid Hormone-related Protein(1-36): Effects on Bone Formation
Brief Title: One Week Parathyroid Hormone-related Protein (PTHrP) IV Dose Escalation Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Mara Horwitz, Associate Professor of Medicne, University of Pittsburgh
Allocation: Non-Randomized | Model: Single Group | Masking: Single
Other Study IDs: PRO07040081; R01DK073039 (NIH)
Record Dates: First submitted 2007-12-20; First posted 2007-12-27 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Osteoporosis; Humoral Hypercalcemia of Malignancy; Hyperparathyroidism
Keywords: Endocrine System Diseases; MusculoSkeletal System Diseases; Hormones; Malignancy; Postmenopausal Women; Bone metabolism
MeSH Terms: conditions — Osteoporosis; Humoral Hypercalcemia Of Malignancy; Hyperparathyroidism; Endocrine System Diseases; Musculoskeletal Diseases; Neoplasms | interventions — parathyroid hormone-related peptide (1-36)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PTHrP(1-36) 2 pmol/kg/hr (Experimental): PTHrP(1-36) at 2 picomoles/kg/hr for one week.
  Interventions: Drug: PTHrP (1-36)
- PTHrP (1-36) 4 pmol/kg/hr (Experimental): PTHrP(1-36) at 4 picomoles/kg/hr for one week.
  Interventions: Drug: PTHrP (1-36)
- PTHrP(1-36) 5 pmol/kg/hr (Experimental): PTHrP(1-36) at 5 picomoles/kg/hr for one week.
  Interventions: Drug: PTHrP (1-36)
- PTHrP(1-36) 6 pmol/kg/hr (Experimental): PTHrP(1-36) at 6 picomoles/kg/hr for one week.
  Interventions: Drug: PTHrP (1-36)

INTERVENTIONS:
Drug: PTHrP (1-36) — IND # 49,175
  Other Names: Parathyroid Hormone-related Protein (1-36)

SUMMARY:
This is a dose escalation study to determine the maximum tolerable dose of Parathyroid Hormone-related Protein, PTHrP, that can be given safely over one week. The investigators plan to infuse low doses of intravenous PTHrP to determine if it leads to a sustained and progressive suppression of bone formation as occurs in humoral hypercalcemia of malignancy (HHM) or an increase in bone formation as occurs in hyperparathyroidism (HPT). Additionally, the investigators will assess the direct influence of PTHrp on markers of bone turnover, and plasma 1,25 (OH)2 vitamin D regulation in healthy human volunteers.

DETAILED DESCRIPTION:
During this research the investigators administer PTHrP to healthy young volunteers in a controlled, continuous intravenous manner. As research subjects complete the week-long study without adverse effects, the dose of PThrP will be increased in later subjects. In the event of a significant adverse effect, immediate action will be taken to reverse it. The investigators want to estimate the effect of a sustainable level of mild hypercalcemia achieved by a week-long intravenous infusion of PTHrP has on vitamin D metabolism, markers of bone turnover and fractional excretion of calcium.

ELIGIBILITY:
Inclusion Criteria:

* Healthy caucasian subjects of both sexes between the ages of 24-35 years, who are able to spend one week on the Clinical & Translational Research Center at the University of Pittsburgh Medical Center (UPMC) Montefiore

Exclusion Criteria:

* Pregnancy
* Any cardiac, renal, pulmonary, endocrine, musculoskeletal, hepatic, hematological, malignant or rheumatologic diseases
* Body mass index great than 30
* Anemia
* Significant alcohol or drug abuse
* Baseline hypotension or hypertension
* Abnormal screening labs
* Use of certain chronic medications excluding oral contraceptives
* Receiving an investigational drug in the last 90 days
* Previously receiving PTH or PTHrP
* African-American race

Ages: 24 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mara J Horwitz, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Juppner H, Abou-Samra AB, Freeman M, Kong XF, Schipani E, Richards J, Kolakowski LF Jr, Hock J, Potts JT Jr, Kronenberg HM, et al. A G protein-linked receptor for parathyroid hormone and parathyroid hormone-related peptide. Science. 1991 Nov 15;254(5034):1024-6. doi: 10.1126/science.1658941.
- [Background] Orloff JJ, Wu TL, Heath HW, Brady TG, Brines ML, Stewart AF. Characterization of canine renal receptors for the parathyroid hormone-like protein associated with humoral hypercalcemia of malignancy. J Biol Chem. 1989 Apr 15;264(11):6097-103. PMID 2539369
- [Background] Orloff JJ, Ribaudo AE, McKee RL, Rosenblatt M, Stewart AF. A pharmacological comparison of parathyroid hormone receptors in human bone and kidney. Endocrinology. 1992 Oct;131(4):1603-11. doi: 10.1210/endo.131.4.1327716.
- [Background] Orloff JJ, Reddy D, de Papp AE, Yang KH, Soifer NE, Stewart AF. Parathyroid hormone-related protein as a prohormone: posttranslational processing and receptor interactions. Endocr Rev. 1994 Feb;15(1):40-60. doi: 10.1210/edrv-15-1-40. PMID 8156938
- [Background] Samuels MH, Veldhuis J, Cawley C, Urban RJ, Luther M, Bauer R, Mundy G. Pulsatile secretion of parathyroid hormone in normal young subjects: assessment by deconvolution analysis. J Clin Endocrinol Metab. 1993 Aug;77(2):399-403. doi: 10.1210/jcem.77.2.8345044.
- [Background] Prank K, Nowlan SJ, Harms HM, Kloppstech M, Brabant G, Hesch RD, Sejnowski TJ. Time series prediction of plasma hormone concentration. Evidence for differences in predictability of parathyroid hormone secretion between osteoporotic patients and normal controls. J Clin Invest. 1995 Jun;95(6):2910-9. doi: 10.1172/JCI117998. PMID 7769133
- [Background] Schmitt CP, Obry J, Feneberg R, Veldhuis JD, Mehls O, Ritz E, Schaefer F. Beta1-adrenergic blockade augments pulsatile PTH secretion in humans. J Am Soc Nephrol. 2003 Dec;14(12):3245-50. doi: 10.1097/01.asn.0000101240.47747.7f. PMID 14638923
- [Background] Chapotot F, Gronfier C, Spiegel K, Luthringer R, Brandenberger G. Relationships between intact parathyroid hormone 24-hour profiles, sleep-wake cycle, and sleep electroencephalographic activity in man. J Clin Endocrinol Metab. 1996 Oct;81(10):3759-65. doi: 10.1210/jcem.81.10.8855835.
- [Background] Harms HM, Schlinke E, Neubauer O, Kayser C, Wustermann PR, Horn R, Kulpmann WR, von zur Muhlen A, Hesch RD. Pulse amplitude and frequency modulation of parathyroid hormone in primary hyperparathyroidism. J Clin Endocrinol Metab. 1994 Jan;78(1):53-7. doi: 10.1210/jcem.78.1.8288713.
- [Background] Ledger GA, Burritt MF, Kao PC, O'Fallon WM, Riggs BL, Khosla S. Role of parathyroid hormone in mediating nocturnal and age-related increases in bone resorption. J Clin Endocrinol Metab. 1995 Nov;80(11):3304-10. doi: 10.1210/jcem.80.11.7593443.
- [Background] el-Hajj Fuleihan G, Klerman EB, Brown EN, Choe Y, Brown EM, Czeisler CA. The parathyroid hormone circadian rhythm is truly endogenous--a general clinical research center study. J Clin Endocrinol Metab. 1997 Jan;82(1):281-6. doi: 10.1210/jcem.82.1.3683. PMID 8989274
- [Background] Plawner LL, Philbrick WM, Burtis WJ, Broadus AE, Stewart AF. Cell type-specific secretion of parathyroid hormone-related protein via the regulated versus the constitutive secretory pathway. J Biol Chem. 1995 Jun 9;270(23):14078-84. doi: 10.1074/jbc.270.23.14078. PMID 7775469
- [Background] Horwitz MJ, Tedesco MB, Sereika SM, Hollis BW, Garcia-Ocana A, Stewart AF. Direct comparison of sustained infusion of human parathyroid hormone-related protein-(1-36) [hPTHrP-(1-36)] versus hPTH-(1-34) on serum calcium, plasma 1,25-dihydroxyvitamin D concentrations, and fractional calcium excretion in healthy human volunteers. J Clin Endocrinol Metab. 2003 Apr;88(4):1603-9. doi: 10.1210/jc.2002-020773. PMID 12679445
- [Background] Syed MA, Horwitz MJ, Tedesco MB, Garcia-Ocana A, Wisniewski SR, Stewart AF. Parathyroid hormone-related protein-(1--36) stimulates renal tubular calcium reabsorption in normal human volunteers: implications for the pathogenesis of humoral hypercalcemia of malignancy. J Clin Endocrinol Metab. 2001 Apr;86(4):1525-31. doi: 10.1210/jcem.86.4.7406. PMID 11297578
- [Background] Everhart-Caye M, Inzucchi SE, Guinness-Henry J, Mitnick MA, Stewart AF. Parathyroid hormone (PTH)-related protein(1-36) is equipotent to PTH(1-34) in humans. J Clin Endocrinol Metab. 1996 Jan;81(1):199-208. doi: 10.1210/jcem.81.1.8550752.
- [Background] Fraher LJ, Hodsman AB, Jonas K, Saunders D, Rose CI, Henderson JE, Hendy GN, Goltzman D. A comparison of the in vivo biochemical responses to exogenous parathyroid hormone-(1-34) [PTH-(1-34)] and PTH-related peptide-(1-34) in man. J Clin Endocrinol Metab. 1992 Aug;75(2):417-23. doi: 10.1210/jcem.75.2.1322424.
- [Background] Horwitz MJ, Tedesco MB, Sereika SM, Syed MA, Garcia-Ocana A, Bisello A, Hollis BW, Rosen CJ, Wysolmerski JJ, Dann P, Gundberg C, Stewart AF. Continuous PTH and PTHrP infusion causes suppression of bone formation and discordant effects on 1,25(OH)2 vitamin D. J Bone Miner Res. 2005 Oct;20(10):1792-803. doi: 10.1359/JBMR.050602. Epub 2005 Jun 6. PMID 16160737
- [Background] Horwitz MJ, Tedesco MB, Sereika SM, Garcia-Ocana A, Bisello A, Hollis BW, Gundberg C, Stewart AF. Safety and tolerability of subcutaneous PTHrP(1-36) in healthy human volunteers: a dose escalation study. Osteoporos Int. 2006 Feb;17(2):225-30. doi: 10.1007/s00198-005-1976-3. Epub 2005 Sep 7. PMID 16151606
- [Background] Plotkin H, Gundberg C, Mitnick M, Stewart AF. Dissociation of bone formation from resorption during 2-week treatment with human parathyroid hormone-related peptide-(1-36) in humans: potential as an anabolic therapy for osteoporosis. J Clin Endocrinol Metab. 1998 Aug;83(8):2786-91. doi: 10.1210/jcem.83.8.5047. PMID 9709948
- [Background] Stewart AF, Mangin M, Wu T, Goumas D, Insogna KL, Burtis WJ, Broadus AE. Synthetic human parathyroid hormone-like protein stimulates bone resorption and causes hypercalcemia in rats. J Clin Invest. 1988 Feb;81(2):596-600. doi: 10.1172/JCI113358. PMID 3339131
- [Background] Burtis WJ, Wu T, Bunch C, Wysolmerski JJ, Insogna KL, Weir EC, Broadus AE, Stewart AF. Identification of a novel 17,000-dalton parathyroid hormone-like adenylate cyclase-stimulating protein from a tumor associated with humoral hypercalcemia of malignancy. J Biol Chem. 1987 May 25;262(15):7151-6. PMID 3584110
- [Background] Stewart AF, Wu T, Goumas D, Burtis WJ, Broadus AE. N-terminal amino acid sequence of two novel tumor-derived adenylate cyclase-stimulating proteins: identification of parathyroid hormone-like and parathyroid hormone-unlike domains. Biochem Biophys Res Commun. 1987 Jul 31;146(2):672-8. doi: 10.1016/0006-291x(87)90581-x. PMID 3619898
- [Background] Wu TL, Vasavada RC, Yang K, Massfelder T, Ganz M, Abbas SK, Care AD, Stewart AF. Structural and physiologic characterization of the mid-region secretory species of parathyroid hormone-related protein. J Biol Chem. 1996 Oct 4;271(40):24371-81. doi: 10.1074/jbc.271.40.24371. PMID 8798692
- [Background] Cosman F, Shen V, Xie F, Seibel M, Ratcliffe A, Lindsay R. Estrogen protection against bone resorbing effects of parathyroid hormone infusion. Assessment by use of biochemical markers. Ann Intern Med. 1993 Mar 1;118(5):337-43. doi: 10.7326/0003-4819-118-5-199303010-00003. PMID 8430979
- [Background] Hodsman AB, Fraher LJ, Ostbye T, Adachi JD, Steer BM. An evaluation of several biochemical markers for bone formation and resorption in a protocol utilizing cyclical parathyroid hormone and calcitonin therapy for osteoporosis. J Clin Invest. 1993 Mar;91(3):1138-48. doi: 10.1172/JCI116273. PMID 8450043
- [Background] Fiaschi-Taesch NM, Stewart AF. Minireview: parathyroid hormone-related protein as an intracrine factor--trafficking mechanisms and functional consequences. Endocrinology. 2003 Feb;144(2):407-11. doi: 10.1210/en.2002-220818. PMID 12538599
- [Derived] Horwitz MJ, Tedesco MB, Sereika SM, Prebehala L, Gundberg CM, Hollis BW, Bisello A, Garcia-Ocana A, Carneiro RM, Stewart AF. A 7-day continuous infusion of PTH or PTHrP suppresses bone formation and uncouples bone turnover. J Bone Miner Res. 2011 Sep;26(9):2287-97. doi: 10.1002/jbmr.415. PMID 21544866

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 subjects were screened and 14 were randomized in the study. Data from 2 subjects was not included in the analysis as there were not enough subjects in that group for analysis. 12 subjects were analyzed.
Groups:
- Group 1: PTHrP(1-36) 2 picomoles/kg/hr
- Group 2: PTHrP(1-36) 4 picomoles/kg/hr
- Group 3: PTHrP (1-36) 5 pmol/kg/hr
- Group 4: PTHrP (1-36) 6 picomoles/kg/hr
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 3 | 6 | 3 | 2
Completed | 3 | 6 | 3 | 1 (One subject was stopped early for hypertension. One subject completed but was not analyzed.)
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 1: PTHrP(1-36) 2 picomoles/kg/hr for one week.
- Group 2: PTHrP(1-36) 4 picomoles/kg/hr for one week.
- Group 3: PTHrP(1-36) 5 picomoles/kg/hr for one week.
- Group 4: PTHrP(1-36) 6 picomoles/kg/hr for one week.
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 3 | 6 | 3 | 2 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 3 | 2 | 14
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 0 | 7
  Male | 1 | 3 | 1 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 3 | 2 | 14

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT)
Description: DLT was defined as achieving one major criterion or two minor criteria rated at ≥ 2 on a scale of 0-5. The major criteria were defined as symptomatic orthostatic hypotension (systolic BP fall >30 mm/hg), tachycardia (pulse > 120), hypertension (systolic BP >160 mm/hg on 2 occasions), hypercalcemia (serum calcium ≥ 12 mg/dl), and hypophosphatemia (serum phosphorous < 1.5 mg/dl). Minor criteria included symptoms such as flushing, nausea, abdominal or muscle cramps, dizziness, lightheadedness, palpitations, etc.
Time Frame: 12 hours after the infusion was started then q 8 hours for 7 days
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 3 | 6 | 3 | 2
participants | 0 | 0 | 2 | 2

2. Secondary Outcome: 1,25 Vitamin D
Description: pg/ml
Time Frame: Baseline and Daily through day 8 then at follow-up visit
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 3 | 6 | 3 | 0
pg/ml
  baseline | 34.13 (3.03) | 45.08 (4.24) | 39.0 (4.09) |
  Day 2 | 38.40 (5.12) | 45.88 (1.53) | 39.77 (2.69) |
  Day 3 | 30.13 (4.57) | 36.58 (4.17) | 36.73 (2.75) |
  Day 4 | 32.23 (2.32) | 40.38 (4.18) | 35.17 (2.63) |
  Day 5 | 32.27 (1.80) | 46.40 (6.12) | 32.07 (3.79) |
  Day 6 | 42.77 (4.23) | 34.90 (4.91) | 35.37 (2.98) |
  Day 7 | 40.53 (4.38) | 37.12 (3.58) | 31.17 (6.84) |
  Day 8 | 32.37 (3.17) | 33.43 (3.13) | 30.63 (4.79) |
  follow-up | 40.10 (4.01) | 45.78 (4.72) | 36.33 (2.11) |
Statistical Analysis 1: Comparison: Group 1 vs Group 3; Test type: Non-Inferiority or Equivalence — The study was designed as a standard dose-escalation study, dose-finding pilot study. The primary outcome measures were safety (hypercalcemia, hypophosphatemia and symptoms/hemodynamic measurements). A modified Fibronacci dose-escalation scheme was employed; p > 0.05, Mixed Models Analysis — The reported p-value corresponds to change over time for the PTHrP 2 and PTHrP 5 pmol groups; The level of statistical significance was set at .05 (two-tailed)
Statistical Analysis 2: Comparison: Group 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.01, Mixed Models Analysis — the reported p value corresponds to a decrease by Day 8 compared to baseline in the PTHrP 4 pmol group; The level of statistical significance was set at .05 (two-tailed)

3. Secondary Outcome: 24 Hour Urine Calcium
Description: mg/gm creatinine collected on day 7 of PTHrP infusion
Time Frame: 24 hours
Measure: Mean (Standard Error); unit: mg/gm creatinine
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 3 | 6 | 3 | 0
mg/gm creatinine | 121.64 (9.87) | 283.43 (30.93) | 320.23 (41.32) |

4. Secondary Outcome: Tubular Maximum of Phosphorous (TmP/GFR)
Description: mg/dl calculated from daily second morning void
Time Frame: daily
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 3 | 6 | 3 | 0
mg/dl
  Baseline | 3.43 (0.26) | 3.91 (0.23) | 3.38 (0.35) |
  Day 2 | 4.48 (0.20) | 4.08 (0.23) | 3.47 (0.46) |
  Day 3 | 4.28 (0.30) | 3.74 (0.26) | 3.25 (0.50) |
  Day 4 | 4.42 (0.31) | 3.75 (0.31) | 3.15 (0.45) |
  Day 5 | 4.43 (0.02) | 3.95 (0.34) | 3.37 (0.45) |
  Day 6 | 4.90 (0.08) | 3.98 (0.11) | 3.38 (0.35) |
  Day 7 | 4.15 (0.08) | 3.98 (0.19) | 2.95 (0.28) |
Statistical Analysis 1: Comparison: Group 1 vs Group 2 vs Group 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.61, Mixed Models Analysis — The reported p-value corresponds to all Arms/Groups at all time points compared to baseline; The level of statistical significance was set at .05 (two-tailed)

5. Primary Outcome: Total Serum Calcium
Description: mg/dl
Time Frame: 12 hours after the infusion was started then q 8 hours for 7 days, Follow-up 1 week after infusion complete
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 3 | 6 | 3 | 0
mg/dl
  baseline | 9.37 (0.07) | 9.58 (0.12) | 9.2 (0.25) |
  11P DAY 1 | 9.67 (0.09) | 9.80 (0.16) | 9.67 (0.20) |
  7A DAY 2 | 9.4 (0.17) | 10.05 (0.19) | 10.17 (0.20) |
  3P DAY 2 | 9.57 (0.09) | 10.28 (0.14) | 10.47 (0.30) |
  11P DAY 2 | 9.67 (0.09) | 10.32 (0.14) | 10.23 (0.26) |
  7A DAY 3 | 9.6 (0.10) | 10.40 (0.18) | 10.73 (0.57) |
  3P DAY 3 | 9.73 (0.09) | 10.42 (0.14) | 10.67 (0.27) |
  11P DAY 3 | 9.40 (0.17) | 9.73 (0.10) | 9.93 (0.38) |
  7A DAY 4 | 9.47 (0.03) | 10.00 (0.24) | 10.3 (0.23) |
  3P DAY 4 | 9.40 (0.17) | 9.92 (0.21) | 10.33 (0.34) |
  11P DAY 4 | 9.37 (0.09) | 9.48 (0.11) | 10.00 (0.15) |
  7A DAY 5 | 9.30 (0.12) | 9.62 (0.12) | 10.53 (0.15) |
  3P DAY 5 | 9.50 (0.15) | 9.83 (0.20) | 10.27 (0.44) |
  11P DAY 5 | 9.43 (0.09) | 9.45 (0.13) | 9.80 (0.20) |
  7A DAY 6 | 9.57 (0.07) | 9.83 (0.20) | 10.53 (0.22) |
  3P DAY 6 | 9.43 (0.15) | 10.08 (0.12) | 10.83 (0.27) |
  11P DAY 6 | 9.43 (0.13) | 9.67 (0.21) | 10.43 (0.47) |
  7A DAY 7 | 9.40 (0.10) | 10.13 (0.28) | 10.90 (0.46) |
  3P DAY 7 | 9.70 (0.15) | 10.22 (0.32) | 10.70 (0.46) |
  11P DAY 7 | 9.60 (0.15) | 10.27 (0.28) | 10.73 (0.50) |
  7A DAY 8 | 9.83 (0.13) | 10.67 (0.40) | 11.17 (0.35) |
  FOLLOW-UP | 9.33 (0.07) | 9.80 (0.12) | 9.17 (0.24) |
Statistical Analysis 1: Comparison: Group 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.0001, Mixed Models Analysis — The reported p-value corresponds to the increase over time for the PTHrP 4 pmol group; Value The level of statistical significance was set at .05 (two-tailed)

6. Primary Outcome: Ionized Serum Calcium
Description: mg/dl
Time Frame: 12 hours after the infusion was started then q 8 hours for 7 days, Follow-up 1 week after infusion complete
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 3 | 6 | 3 | 0
mg/dl
  baseline | 4.79 (0.03) | 4.72 (0.08) | 4.55 (0.15) |
  11P DAY 1 | 4.51 (0.05) | 4.77 (0.08) | 4.75 (0.04) |
  7A DAY 2 | 4.77 (0.07) | 4.98 (0.10) | 5.07 (0.07) |
  3P DAY 2 | 4.52 (0.02) | 4.99 (0.06) | 5.07 (0.06) |
  11P DAY 2 | 4.48 (0.08) | 5.04 (0.07) | 4.84 (0.00) |
  7A DAY 3 | 4.77 (0.15) | 5.31 (0.08) | 5.25 (0.13) |
  3P DAY 3 | 4.73 (0.11) | 4.99 (0.10) | 4.91 (0.16) |
  11P DAY 3 | 4.41 (0.15) | 4.58 (0.15) | 4.83 (0.14) |
  7A DAY 4 | 4.75 (0.14) | 4.90 (0.13) | 5.11 (0.09) |
  3P DAY 4 | 4.45 (0.16) | 4.68 (0.14) | 4.72 (0.17) |
  11P DAY 4 | 4.47 (0.07) | 4.46 (0.12) | 4.69 (0.06) |
  7A DAY 5 | 4.71 (0.07) | 4.82 (0.09) | 4.97 (0.12) |
  3P DAY 5 | 4.61 (0.20) | 4.67 (0.12) | 4.87 (0.40) |
  11P DAY 5 | 4.60 (0.13) | 4.58 (0.07) | 4.79 (0.09) |
  7A DAY 6 | 4.63 (0.03) | 4.77 (0.10) | 5.25 (0.09) |
  3P DAY 6 | 4.72 (0.13) | 4.83 (0.07) | 5.35 (0.03) |
  11P DAY 6 | 4.32 (0.06) | 4.72 (0.09) | 5.19 (0.21) |
  7A DAY 7 | 4.55 (0.22) | 5.01 (0.09) | 5.55 (0.27) |
  3P DAY 7 | 4.84 (0.16) | 5.04 (0.17) | 5.25 (0.31) |
  11P DAY 7 | 4.56 (0.12) | 4.87 (0.19) | 5.24 (0.02) |
  7A DAY 8 | 5.00 (0.11) | 5.43 (0.18) | 5.69 (0.10) |
  FOLLOW-UP | 4.68 (0.08) | 4.83 (0.05) | 4.80 (0.06) |
Statistical Analysis 1: Comparison: Group 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.0001, Mixed Models Analysis — The reported p-value corresponds to the increase over time for the PTHrP 4 pmol group; The level of statistical significance was set at .05 (two-tailed)

7. Primary Outcome: Serum Phosphorous
Description: mg/dl
Time Frame: 12 hours after the infusion was started then q 8 hours for 7 days, Follow-up 1 week after infusion complete
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 3 | 6 | 3 | 0
mg/dl
  baseline | 3.55 (0.15) | 3.63 (0.14) | 3.55 (0.45) |
  11P DAY 1 | 3.87 (0.26) | 3.90 (0.16) | 4.03 (0.12) |
  7A DAY 2 | 4.07 (0.15) | 4.20 (0.15) | 3.63 (0.44) |
  3P DAY 2 | 3.63 (0.33) | 3.50 (0.23) | 3.70 (0.20) |
  11P DAY 2 | 4.13 (0.29) | 3.52 (0.19) | 3.63 (0.19) |
  7A DAY 3 | 3.90 (0.26) | 3.77 (0.19) | 3.43 (0.39) |
  3P DAY 3 | 3.53 (0.24) | 3.53 (0.18) | 3.60 (0.23) |
  11P DAY 3 | 4.03 (0.26) | 3.58 (0.17) | 3.70 (0.15) |
  7A DAY 4 | 4.07 (0.22) | 3.90 (0.13) | 3.30 (0.40) |
  3P DAY 4 | 3.90 (0.10) | 3.37 (0.20) | 3.33 (0.32) |
  11P DAY 4 | 3.67 (0.28) | 3.48 (0.14) | 3.63 (0.27) |
  7A DAY 5 | 3.87 (0.19) | 4.02 (0.14) | 3.20 (0.30) |
  3P DAY 5 | 3.57 (0.29) | 3.35 (0.20) | 3.10 (0.21) |
  11P DAY 5 | 3.93 (0.23) | 3.45 (0.20) | 3.87 (0.32) |
  7A DAY 6 | 4.00 (0.06) | 4.00 (0.10) | 3.63 (0.35) |
  3P DAY 6 | 3.67 (0.03) | 3.80 (0.14) | 3.73 (0.19) |
  11P DAY 6 | 3.93 (0.18) | 3.90 (0.10) | 3.93 (0.09) |
  7A DAY 7 | 4.30 (0.10) | 4.28 (0.12) | 3.73 (0.38) |
  3P DAY 7 | 4.07 (0.09) | 3.62 (0.20) | 3.50 (0.20) |
  11P DAY 7 | 4.20 (0.26) | 3.62 (0.19) | 3.60 (0.30) |
  7A DAY 8 | 4.43 (0.15) | 4.10 (0.10) | 3.40 (0.23) |
  FOLLOW-UP | 3.57 (0.38) | 3.48 (0.26) | 3.87 (0.09) |
Statistical Analysis 1: Comparison: Group 1 vs Group 2 vs Group 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p > .05, Mixed Models Analysis — The reported p-value corresponds to change over time from baseline for all Arms/groups; The level of statistical significance was set at .05 (two-tailed)

8. Secondary Outcome: Serum Amino-terminal Telopeptide of Collagen -1 (sNTX)
Description: % change from baseline
Time Frame: Baseline, Daily, and 1 week follow-up
Measure: Mean (Standard Error); unit: % change
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 3 | 6 | 3 | 0
% change
  baseline | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) |
  Day 2 | 32.86 (23.41) | 87.75 (18.79) | 54.21 (10.64) |
  Day 3 | 26.73 (23.19) | 91.53 (28.94) | 88.51 (19.99) |
  Day 4 | 28.32 (20.26) | 90.86 (32.25) | 89.57 (20.22) |
  Day 5 | 41.29 (20.06) | 82.36 (20.62) | 116.58 (13.85) |
  Day 6 | 11.41 (12.63) | 123.08 (28.62) | 150.82 (48.26) |
  Day 7 | 35.04 (21.44) | 161.55 (41.54) | 176.42 (50.08) |
  Day 8 | 65.77 (30.43) | 214.90 (59.26) | 108.69 (34.29) |
  follow-up | -14.95 (2.97) | -3.33 (6.68) | -9.02 (7.19) |
Statistical Analysis 1: Comparison: Group 1 vs Group 2 vs Group 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < .008, Mixed Models Analysis — The reported p-value corresponds to the % increase compared to baseline in all Arms/groups on Days 2-8; The level of statistical significance was set at .05 (two-tailed)
Statistical Analysis 2: Comparison: Group 1 vs Group 2 vs Group 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p > 0.05, Mixed Models Analysis — The reported p-value corresponds the the % change from baseline at follow-up in all Arms/groups; The level of statistical significance was set at .05 (two-tailed)

9. Secondary Outcome: Serum Carboxy-terminal Telopeptide of Collagen -1 (sCTX)
Description: % change from baseline
Time Frame: Baseline, Daily, and 1 week follow-up
Measure: Mean (Standard Error); unit: % change
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 3 | 6 | 3 | 0
% change
  baseline | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) |
  Day 2 | 59.78 (18.14) | 147.12 (40.72) | 105.06 (11.54) |
  Day 3 | 66.67 (32.24) | 180.27 (44.45) | 148.45 (36.80) |
  Day 4 | 71.19 (18.88) | 167.01 (47.01) | 165.16 (40.29) |
  Day 5 | 79.39 (23.89) | 167.27 (25.30) | 174.58 (47.26) |
  Day 6 | 74.09 (26.72) | 239.51 (49.42) | 230.42 (54.10) |
  Day 7 | 109.27 (29.39) | 283.15 (65.65) | 267.89 (104.52) |
  Day 8 | 110.61 (30.92) | 368.31 (93.63) | 140.58 (78.58) |
  follow-up | -35.73 (11.53) | -8.60 (11.15) | -41.33 (20.38) |
Statistical Analysis 1: Comparison: Group 1 vs Group 2 vs Group 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < .0001, Mixed Models Analysis — The reported p-value corresponds to % change (increase) from baseline in all Arms/groups at Days 2-8; The level of statistical significance was set at .05 (two-tailed)
Statistical Analysis 2: Comparison: Group 1 vs Group 2 vs Group 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p > 0.05, Mixed Models Analysis — The reported p-value corresponds to the % change from baseline at follow-up in all Arms/groups; The level of statistical significance was set at .05 (two-tailed)

10. Secondary Outcome: Amino-terminal Peptides of Procollagen 1 (P1NP)
Description: % change from baseline
Time Frame: Baseline, Daily, and 1 week follow-up
Measure: Mean (Standard Error); unit: % change
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 3 | 6 | 3 | 0
% change
  baseline | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) |
  Day 2 | -1.05 (4.95) | -17.49 (5.93) | -23.88 (6.05) |
  Day 3 | -6.83 (2.78) | -30.44 (7.10) | -37.77 (6.56) |
  Day 4 | -12.16 (0.57) | -25.66 (9.55) | -39.44 (4.46) |
  Day 5 | -5.63 (2.27) | -21.27 (8.01) | -45.04 (3.07) |
  Day 6 | -8.42 (5.07) | -31.71 (7.50) | -39.55 (1.75) |
  Day 7 | -12.59 (6.17) | -30.98 (8.87) | -39.88 (2.78) |
  Day 8 | -16.03 (5.03) | -36.60 (9.64) | -38.53 (3.40) |
  follow-up | -7.12 (2.29) | 0.60 (9.58) | 46.67 (17.34) |
Statistical Analysis 1: Comparison: Group 1 vs Group 2 vs Group 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < .0001, Mixed Models Analysis — the reported p-value corresponds to % decrease compared to baseline at Days 2-8 in all Arms/groups; The level of statistical significance was set at .05 (two-tailed)
Statistical Analysis 2: Comparison: Group 1 vs Group 2 vs Group 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.01, Mixed Models Analysis — the reported p-value corresponds to % change from baseline at the follow-up visit in all Arms/groups; The level of statistical significance was set at .05 (two-tailed)

11. Secondary Outcome: Bone Specific Alkaline Phosphatase (BSAP)
Description: % change from baseline
Time Frame: Baseline, Daily, and 1 week follow-up
Measure: Mean (Standard Error); unit: % change
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 3 | 6 | 3 | 0
% change
  baseline | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) |
  Day 2 | -12.53 (8.60) | -1.17 (4.10) | 24.54 (7.01) |
  Day 3 | -6.35 (4.84) | -1.44 (3.07) | 34.77 (6.53) |
  Day 4 | -5.82 (1.58) | -3.79 (4.65) | 19.49 (8.23) |
  Day 5 | -0.33 (0.33) | -9.64 (4.73) | 13.61 (9.76) |
  Day 6 | -8.16 (9.32) | -10.88 (4.04) | 9.02 (8.94) |
  Day 7 | -11.91 (10.38) | -16.78 (2.58) | 9.86 (4.01) |
  Day 8 | -7.80 (8.66) | -14.01 (3.72) | 15.27 (11.63) |
  follow-up | -1.25 (2.70) | 6.16 (3.81) | 18.23 (2.22) |
Statistical Analysis 1: Comparison: Group 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.001, Mixed Models Analysis — the reported p-value correspond to the decrease compared to baseline over time in the PTHrP 4 pmol group; The level of statistical significance was set at .05 (two-tailed)
Statistical Analysis 2: Comparison: Group 1 vs Group 2 vs Group 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = .01, Mixed Models Analysis — the reported p=value corresponds to % change compared to baseline at follow-up in all Arms/groups; The level of statistical significance was set at .05 (two-tailed)

12. Secondary Outcome: Parathyroid Hormone (1-84)
Description: pg/ml
Time Frame: Baseline and Daily
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 3 | 6 | 3 | 0
pg/ml
  baseline | 42.97 (2.86) | 30.70 (5.56) | 48.27 (15.93) |
  Day 2 | 23.47 (1.48) | 7.82 (1.50) | 3.60 (0.50) |
  Day 3 | 21.43 (3.65) | 5.23 (1.75) | 3.00 (0.00) |
  Day 4 | 26.77 (3.24) | 7.88 (3.21) | 3.00 (0.00) |
  Day 5 | 22.37 (5.10) | 7.54 (1.80) | 3.00 (0.00) |
  Day 6 | 21.13 (5.88) | 6.57 (2.24) | 3.00 (0.00) |
  Day 7 | 19.40 (4.03) | 5.67 (1.20) | 3.00 (0.00) |
  Day 8 | 12.60 (3.58) | 3.00 (0.00) | 3.00 (0.00) |
  follow-up | 56.37 (5.18) | 31.60 (2.63) | 44.20 (10.87) |
Statistical Analysis 1: Comparison: Group 1 vs Group 2 vs Group 3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.05, Mixed Models Analysis — the reported p-values correspond to the decrease compared to baseline in all arms/groups at Days 2-8; The level of statistical significance was set at .05 (two-tailed)

13. Secondary Outcome: Fractional Excretion of Calcium
Description: % calculated from daily second morning void
Time Frame: daily
Measure: Mean (Standard Error); unit: % of filtered load
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 3 | 6 | 3 | 0
% of filtered load
  Baseline | 1.93 (0.91) | 2.57 (0.73) | 2.38 (0.59) |
  Day 2 | 1.31 (0.59) | 2.26 (0.46) | 4.11 (2.42) |
  Day 3 | 1.07 (0.51) | 2.85 (0.61) | 3.27 (0.45) |
  Day 4 | 1.57 (0.25) | 2.79 (0.76) | 2.14 (0.40) |
  Day 5 | 3.05 (0.70) | 2.05 (0.46) | 3.12 (0.46) |
  Day 6 | 3.37 (0.67) | 2.75 (0.25) | 5.42 (2.23) |
  Day 7 | 2.72 (0.28) | 3.94 (0.38) | 4.13 (0.73) |
Statistical Analysis 1: Comparison: Group 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p = .002, Mixed Models Analysis — the reported p-value corresponds to the increase comapred to baseline over time (days 2-8) in the PTHrP 4 pmol group; The level of statistical significance was set at .05 (two-tailed)

ADVERSE EVENTS:
Time Frame: Subjects were systematically assessed every 8 hours for adverse events
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 1/3 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=3) | Group 2 (N=6) | Group 3 (N=3) | Group 4 (N=2)
hypercalcemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
hypertension (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
migraine (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
lightheaded (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
tachycardia (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small number of subjects in each group Study limited to Caucasians Only one timepoint for follow-up was measure Study did not include saline infused controls

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No